CLINICAL TRIAL: NCT01599520
Title: Stress Management Training for Latinas Receiving Chemotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCC-16956
Record Dates: First submitted 2012-04-23; First posted 2012-05-16 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Cancer; Stress
Keywords: cancer; stress; stress management; Latinas; Hispanics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spanish-Language Self-Administered Training + Usual Care (Experimental): Participants randomized to this arm will receive Spanish-Language Self-Administered Training + Usual Care.
  Interventions: Behavioral: Spanish-Language Self-Administered Training Plus Usual Care (SL-SAT)
- Usual Care Only (Active Comparator): Patients will be given the Spanish-language version of "Chemotherapy and You: Support for People with Cancer" ("La quimioterapia y usted: Apoyo para las personas con cancer") published by NCI. The intervention associate will review how it provides answers to common questions about chemotherapy, describes common side effects and their management, and identifies ways to obtain additional information. Patients will also be provided with a list of local support groups for cancer patients and informed that a social worker is available to meet with them without charge to discuss personal concerns or practical problems. At the first infusion, oncology nurses will provide all patients with standard education about the chemotherapy agents and anti-emetic agents to be administered, possible adverse reactions to these agents, and recommended precautions for avoiding illness and maintaining health.
  Interventions: Behavioral: Usual Care Only

INTERVENTIONS:
Behavioral: Spanish-Language Self-Administered Training Plus Usual Care (SL-SAT) — Patients will receive usual care. In addition, a Spanish-speaking intervention associate will spend an extra 10 minutes on the day usual care is initiated reviewing the self-administered training materials in Spanish titled "Cómo tratar el estrés durante la quimioterapia." Materials consist of an 18-minute DVD (also available as a videocassette (VC)), a 28-minute CD (also available as an audiocassette (AC)), a 16-page booklet, and a workbook to record practice and use of stress management techniques. Participants are instructed to first view the DVD/VC and then follow directions in the booklet and on the CD/AC about training, practice, and use of stress management techniques.
  Arms: Spanish-Language Self-Administered Training + Usual Care
Behavioral: Usual Care Only — Patients will be given the Spanish-language version of "Chemotherapy and You: Support for People with Cancer" ("La quimioterapia y usted: Apoyo para las personas con cancer") published by NCI. The intervention associate will review how it provides answers to common questions about chemotherapy, describes common side effects and their management, and identifies ways to obtain additional information. Patients will also be provided with a list of local support groups for cancer patients and informed that a social worker is available to meet with them without charge to discuss personal concerns or practical problems. At the first infusion, oncology nurses will provide all patients with standard education about the chemotherapy agents and anti-emetic agents to be administered, possible adverse reactions to these agents, and recommended precautions for avoiding illness and maintaining health.
  Arms: Usual Care Only

SUMMARY:
Cancer patients receiving chemotherapy experience a number of aversive symptoms that are accompanied by declines in physical and mental well-being. Although the benefits of stress management training interventions on quality of life are well documented, there are no published studies examining the efficacy of these interventions among Hispanic women and Latinas (hereafter referred to as Latinas) receiving chemotherapy. This dearth of research reflects the general lack of stress management interventions for cancer patients whose preferred language is Spanish. Simply translating existing English-language interventions into Spanish may seem to be a solution for the lack of Spanish-language stress management interventions. This approach, however, does not take into account cultural values, beliefs and situational realities that are likely to contribute to patients' uptake of health promoting behaviors. The proposed research seeks to address this gap by evaluating a stress management training intervention developed specifically for Latinas beginning chemotherapy for cancer.

In response to the identified need, the investigators created a Spanish-Language Self-Administered Stress Management Training (SL-SAT) intervention "Cómo tratar el estrés durante la quimioterapia" ("How to manage stress during chemotherapy"). The intervention is based on an English-language self-administered stress management training intervention the investigators previously developed and showed to be efficacious in a randomized controlled trial. Development of the Spanish-language intervention was the result of extensive use of ethnographic and learner verification methods, guided by a community-based participatory research approach. Similar to the English-language version, the SL-SAT intervention consists of a digital video disc(DVD), booklet, and audio compact disc (CD), and provides instruction in three well-established stress management techniques: deep breathing; progressive muscle relaxation and guided imagery; and use of coping self-statements. The proposed study will evaluate the efficacy of this transcreated intervention in a randomized controlled trial involving Spanish-speaking Latinas about to begin chemotherapy for cancer. Following a baseline assessment, participants will receive usual care or usual care plus the SL-SAT intervention. Participants will be reassessed on study measures approximately 7 and 13 weeks after the baseline assessment.

DETAILED DESCRIPTION:
Specific aims of the project are:

1. To evaluate the impact of Cómo tratar el estrés durante la quimioterapia on quality of life during chemotherapy relative to usual care only. Consistent with prior research, the investigators hypothesize that the intervention will result in better psychological and spiritual well-being and less anxiety, depression, and cancer-related distress.
2. To investigate the mechanism by which Cómo tratar el estrés durante la quimioterapia improves quality of life during chemotherapy. Based on relevant theory and prior research, the investigators hypothesize that improvement in perceived self-efficacy in managing stress will explain beneficial effects of the intervention on quality of life outcomes.
3. To examine whether communication and sociocultural factors associated with the acculturation process moderate the impact of Cómo tratar el estrés durante la quimioterapia on quality of life. Based on relevant theory and prior research, the investigators hypothesize that, among women who receive the intervention, those who have a stronger preference for communicating and receiving information in Spanish will benefit more.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be female
* Self-identify as Hispanic or Latina
* Be capable of speaking and reading Spanish
* Be diagnosed with cancer
* Be scheduled to start outpatient intravenous (IV) chemotherapy for reasons other than symptom palliation at Moffitt Cancer Center (MCC)
* Be scheduled to receive chemotherapy on one of the five schedules specified in Table 3
* Have not received chemotherapy in the past 2 months
* Have no documented or observable visual, auditory, psychiatric, or neurological disorders that would interfere with participation (e.g., blindness, deafness, psychosis, or dementia)
* Be able to provide written informed consent

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2012-03-13 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2021-11-19 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale (HADS) | Baseline, Week 5-7, Week 13 (to evaluate change)
  This 14-item measure has been used widely in behavioral oncology research because it does not assess somatic symptoms of anxiety and depression (e.g., fatigue) that may be confounded with disease- or treatment-related symptoms. The validated Spanish version will be used in the current study. Analyses will focus on the total score as a primary outcome.
Impact of Event-Revised Intrusion Subscale (IES-R) | Baseline, Week 5-7, Week 13 (to evaluate change)
  The 8-item Intrusion Subscale from the IES-R measures intrusive thoughts, such as dreams, images, and reminders of a stressful event. In the present study, as in other research, it will be keyed to "your cancer and cancer diagnosis" in order to provide a measure of cancer-related distress. The IES-R has been validated in numerous populations and is widely used in cancer research. The validated Spanish version will be used in the current study.
Functional Assessment of Cancer Therapy--General Version | Baseline, 5-7 weeks, 13 weeks (to evaluate change)
  This 27-item measure has been used to assess health-related quality of life in patients with many different types of cancer. The validated Spanish version will be used in the current study.The FACT-G yields scores for physical, social/family, emotional, and functional well-being. Analyses will focus on emotional well-being scores as a primary outcome; other scales will be examined as secondary outcomes.
Functional Assessment of Chronic Illness-Spiritual Well-being Scale (FACIT-SP) | Baseline, 5-7 weeks, 13 weeks (to evaluate change)
  This 12-item scale is a valid and reliable measure of spiritual well-being in cancer patients. The validated Spanish version will be used in the current study. The FACIT-Sp yields scores for meaning/peace and faith as well as a total score. Analyses will focus on total FACIT-Sp scores as a primary outcome.

SECONDARY OUTCOMES:
Memorial Symptom Assessment Scale-Short Form (MSAS-SF) | Baseline, 5-7 weeks, 13 weeks
  This scale is a valid and reliable measure of the severity of 32 symptoms commonly experienced by cancer patients (e.g., nausea, vomiting, and lack of appetite). The Spanish version produced by the original scale developers will be used in the current study. Responses yield measures of the severity of individual symptoms that can also be combined to yield indices of total, physical, and psychological symptom severity. MSAS-SF summary scale scores will be examined as secondary outcomes in the current study.
Measure of Current Status (MOCS) | Baseline, 5-7 weeks, 13 weeks
  This 17-item measure assesses perceived self-efficacy in managing stress. Items closely mirror stress management strategies that comprise the SL-SAT intervention. Based on our conceptual model and previous research with cancer patients, the investigators will examine whether perceived self-efficacy, as measured by the MOCS, mediates the expected positive effects of the SL-SAT intervention on the primary outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Brian D Gonzalez, Ph.D, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States